CLINICAL TRIAL: NCT06650657
Title: The Effect of Touchpoint Method on Clinical Learning
Brief Title: The Effect of Touchpoint Method on Clinical Learning; Experience With Nursing Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Yasemin Ciraci Yasar, primary author, Ataturk University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ATATURKU-NRS-YCY-03
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Educational Problems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): touchpoint method
  Interventions: Behavioral: touchpoint method
- Arm 2 (No Intervention): usual learning method

INTERVENTIONS:
Behavioral: touchpoint method — Touchpoint is a quality approach that can be applied to increase the sense of personal connection with the instructor, ensure that students are making satisfactory progress, increase instructor-student and student-instructor interactions, and increase student satisfaction, unlike traditional learning models.
  Arms: Arm 1

SUMMARY:
This research aims to evaluate the effect of Touchpoint experience as a clinical learning method on clinical learning. The research is a quasi-experimental research with experimental-control groups. Students will be divided into experimental and control groups with the "simple randomization" method. A pre-test will be taken with data collection tools before the study for both groups. Students in the control group will continue their routine practice experiences. A post-test will be applied with data collection tools at the end of the 8-week internship period. TouchPoint is planned as a 2-session experience over a semester: Session 1 focuses on patient-centered care, Session 2 focuses on teamwork and collaboration. The method of both sessions will be conducted by 2 researchers with a small clinical group of 8 to 10 students. Sessions will last from 1.5 hours to 2 hours depending on the number of students and the degree of discussion. Sessions will be conducted face-to-face in a classroom.

DETAILED DESCRIPTION:
Outcome Measures:

Clinical Learning Climate Scale: This measurement tool used in the study was developed by Demiral Yılmaz (2010). This scale consists of 36 items (Demir Yılmaz, 2010). The scale is scored using a 5-point Likert scale (I completely disagree: 1 - I completely agree: 5). Three dimensions are defined in the factor analysis of the scale. These dimensions are; clinical environment, emotional climate and motivation.

Student Satisfaction Scale-Short Form: SSS-SF is the shortened and revised version of the "Student Satisfaction Scale" developed by Baykal et al. to determine the satisfaction of students studying at nursing schools, by Baykal et al. in 2011. In the evaluation of the 53 items in the scale, a five-point Likert-type measurement is used, including "5-Strongly agree, 4- Agree, 3-Undecided, 2-Disagree, 1-Strongly disagree". As the average score approaches 1 in the scale as a whole and in the sub-dimensions, the student is considered to be dissatisfied, and as the score approaches 5, the student is considered to be satisfied. The scale was found to be highly reliable, with a Cronbach's alpha coefficient of 0.97 in total. The scale has 5 sub-dimensions, namely, faculty members, school administration, participation in decisions, scientific, social and technical opportunities, and quality of education. The highest score that can be obtained from the scale is 265 and the lowest score is 53. As the average score on the scale as a whole and in the sub-dimensions approaches 1, the student is considered to be insatiable, and as the score approaches 5, the student is considered to be satisfied.

Eligibility Criteria: Being a 2nd year student at the Faculty of Nursing, Agreeing to participate in the research

ELIGIBILITY:
Inclusion Criteria:

* Being a 2nd year student at the Faculty of Nursing,
* Agreeing to participate in the research

Exclusion Criteria:

* Not being a 2nd year student at the Faculty of Nursing,
* Not agreeing to participate in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Learning Climate Scale | 8 weeks
  This scale consists of 36 items The scale is scored using a 5-point Likert scale (I completely disagree: 1 - I completely agree: 5). Three dimensions are defined in the factor analysis of the scale. These dimensions are; clinical environment, emotional climate and motivation.
Student Satisfaction Scale-Short Form | 8 weeks
  In the evaluation of the 53 items in the scale, a five-point Likert-type measurement is used, including "5-Strongly agree, 4- Agree, 3-Undecided, 2-Disagree, 1-Strongly disagree". As the average score approaches 1 in the scale as a whole and in the sub-dimensions, the student is considered to be dissatisfied, and as the score approaches 5, the student is considered to be satisfied. The scale was found to be highly reliable, with a Cronbach's alpha coefficient of 0.97 in total. The scale has 5 sub-dimensions, namely, faculty members, school administration, participation in decisions, scientific, social and technical opportunities, and quality of education. The highest score that can be obtained from the scale is 265 and the lowest score is 53. As the average score on the scale as a whole and in the sub-dimensions approaches 1, the student is considered to be insatiable, and as the score approaches 5, the student is considered to be satisfied.

IPD SHARING:
Plan to Share IPD: No